CLINICAL TRIAL: NCT00457457
Title: A Multi-center, Randomized, Parallel Group, Double-blind, Placebo Controlled Proof of Concept and Dose Ranging Study With an Active Control to Assess the Efficacy and Safety/Tolerability of UK-369,003 Immediate Release (IR) and Modified Release (MR) in the Treatment of Men With Lower Urinary Tract Symptoms (LUTS) With and Without Erectile Dysfunction (ED)
Brief Title: Study the Effects of Different Doses of UK-369,003 in Men With Lower Urinary Tract Symptoms.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3711044
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Prostatic Hyperplasia
Keywords: With or without erectile dysfunction
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin; 1-(6-ethoxy-5-(3-ethyl-6,7-dihydro-2-(2-methoxyethyl)-7-oxo-2H-pyrazolo(4,3-d)pyrimidin-5-yl)-3-pyridyl sulphonyl)-4-ethylpiperazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparator (Active Comparator): Tamsulosin 0.4 mg prolonged release
  Interventions: Drug: Tamsulosin
- Treatment Arm (Experimental): There are 5 possible UK-369,003 arms as follows: UK-369,003 MR (10mg, 25mg, 50mg & 100mg), UK-369,003 IR (40mg),
  Interventions: Drug: UK-369,003

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin hydrochloride capsules, 0.4 mg. Tamsulosin hydrochloride is an antagonist of alpha1A adrenoceptors in the prostate
  Arms: Comparator
Drug: UK-369,003 — UK 369,003 is a highly selective and potent inhibitor of PDE5. It has increased selectivity for PDE5 over PDE6 (>80 fold) compared to sildenafil (~10 fold). Two recently completed trials have shown efficacy for UK-369,003 in treating subjects with ED
  Arms: Treatment Arm

SUMMARY:
This is a 12 week study in which different doses and formulations of UK-369,003 will be administered to patients with a diagnosis of enlarged prostate. Patients will complete a series of questionnaires before, during and after treatment to assess if UK-369,003 has improved their urinary symptoms and erectile function . There will be several blood samples taken during the study to asses the level of drug in the blood and correlate it with the responses to the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged 40 years and above, with documented LUTS with an International Prostate Symptom Score (IPSS) ≥13
2. Clinical diagnosis of BPH.
3. Qmax 5 to 15ml/sec with a voided volume of ≥150ml at visit 1 (screening).

Exclusion Criteria:

1. Urinary tract infection
2. Primary neurological conditions affecting bladder function

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change in international prostate symptom score | 12 weeks

SECONDARY OUTCOMES:
Erectile Function (EF) domain of International Index of Erectile | 12 weeks
Function (IIEF) | 12 weeks
Qmax | 12 weeks
Quality of Erection questionnaire (QEQ) | 12 weeks
Population pharmacokinetics | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- Australia (2):
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
- Canada (3):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Pointe-Claire, Quebec
- Chile (2):
  - Pfizer Investigational Site, Temuco, Región de la Araucanía
  - Pfizer Investigational Site, Santiago
- Colombia (4):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Cali, Valle del Cauca Department
- Denmark (3):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Aarhus N
  - Pfizer Investigational Site, Gentofte Municipality
- Finland (4):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Oulu
  - Pfizer Investigational Site, Tampere
- Greece (3):
  - Pfizer Investigational Site, Larissa
  - Pfizer Investigational Site, Rio
  - Pfizer Investigational Site, Thessaloniki
- Italy (2):
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Siena
- Pfizer Investigational Site, Riga, Latvia
- Lithuania (2):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Vilnius
- Poland (5):
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Gdynia
  - Pfizer Investigational Site, Mysłowice
  - Pfizer Investigational Site, Wejherowo
- Slovakia (5):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Malacky
  - Pfizer Investigational Site, Nitra
  - Pfizer Investigational Site, Prešov
  - Pfizer Investigational Site, Skalica
- Spain (3):
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Málaga
  - Pfizer Investigational Site, Valencia
- Pfizer Investigational Site, Bristol, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3711044&StudyName=Study%20the%20effects%20of%20different%20doses%20of%20UK-369%2C003%20in%20men%20with%20lower%20urinary%20tract%20symptoms.%20%20